CLINICAL TRIAL: NCT03587493
Title: Activated Cytotoxic T-lymphocytes CD8+/HLA-DR+ and Acute Cellular Rejection After Lung Transplantation
Brief Title: T-lymphocytes CD8+/HLA-DR+ and Acute Rejection After Lung Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-09
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Transplant Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXPERIMENTAL GROUP (Experimental): 110 adults, on national waiting list for a first lung transplantation in the centers of Marseille and Strasbourg, whatever the lung disease, and who will be transplanted and benefit immunosuppressive induction therapy that specifically targets T lymphocytes will be included.
  Blood sample analysis will be performed
  Interventions: Other: BLOOD SAMPLE ANALYSIS

INTERVENTIONS:
Other: BLOOD SAMPLE ANALYSIS — Peripheral venous blood sampling just before lung transplantation, at day 15 and at post-transplantation M1 for lymphocyte phenotyping by cytometry

SUMMARY:
The objectives of the study is to identify associations between acute rejection and the increase of T (CD4/CD8) and B circulating lymphocytes expressing specific markers of activation and differentiation (HLA-DR, CD25, CD38, CD45RO, CCR7).

110 adults over 18 years, on national waiting list for a first lung transplantation in the centers of Marseille and Strasbourg, whatever the lung disease, and who will be transplanted and benefit immunosuppressive induction therapy that specifically targets T lymphocytes will be included. Peripheral venous blood sampling just prior to pulmonary transplantation, at day 15 and one month post-transplant will be realized for lymphocyte phenotyping by flow cytometry (CD45, CD3, CD4, CD8, CD19, HLA-DR, CD25, CD38, CD45RO, CCR7). Acute rejection will be evaluated at 1 month and 1 year post-transplant by trans-bronchial biopsies.

The two main perspectives are to 1) find a specific, non-invasive, blood-based diagnostic marker of acute post-lung transplant rejection with diagnostic performance equivalent to trans-bronchial biopsy 2) demonstrate a specific blood marker, non-invasive, predictive of acute rejection in order to adapt immunosuppressive therapy early and reduce the occurrence of this risk.

DETAILED DESCRIPTION:
The objectives of the study is to identify associations between acute rejection and the increase of T (CD4/CD8) and B circulating lymphocytes expressing specific markers of activation and differentiation (HLA-DR, CD25, CD38, CD45RO, CCR7).

110 adults over 18 years, on national waiting list for a first lung transplantation in the centers of Marseille and Strasbourg (France), whatever the lung disease, and who will be transplanted and benefit immunosuppressive induction therapy that specifically targets T lymphocytes will be included. Peripheral venous blood sampling just prior to pulmonary transplantation, at day 15 and one month post-transplant will be realized for lymphocyte phenotyping by flow cytometry (CD45, CD3, CD4, CD8, CD19, HLA-DR, CD25, CD38, CD45RO, CCR7). Acute rejection will be evaluated at 1 month and 1 year post-transplant by trans-bronchial biopsies.

The two main perspectives are to 1) find a specific, non-invasive, blood-based diagnostic marker of acute post-lung transplant rejection with diagnostic performance equivalent to trans-bronchial biopsy 2) demonstrate a specific blood marker, non-invasive, predictive of acute rejection in order to adapt immunosuppressive therapy early and reduce the occurrence of this risk.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* French national waiting list of lung transplantation
* Transplanted in Marseille or Strasbourg (France)

Exclusion Criteria:

* <18 years old
* Refused to participate
* Redo lung transplantation
* Other organ transplanted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
T-lymphocytes CD8/HLA-DR+ | at day 15 post lung transplantation
  comparison of the level of T-lymphocytes CD8/HLA-DR+ at day 15 post lung transplantation between recipients who developed acute cellular rejection at 1 month post-transplant and those who not.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France